CLINICAL TRIAL: NCT06564324
Title: A Phase 3 Multicenter Open-label Study of Taletrectinib Versus a Standard of Care ROS1-Tyrosine Kinase Inhibitor (Crizotinib) in TKI-Naïve Patients With ROS1-Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer (TRUST-III)
Brief Title: A Phase III Study Comparing Taletrectinib With Standard Therapy in ROS1 Positive Locally Advanced or Metastatic Non-small Cell Lung Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nuvation Bio Inc. (Industry)
Collaborators: AnHeart Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB-106-G318
Record Dates: First submitted 2024-08-12; First posted 2024-08-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — taletrectinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taletrectinib (Experimental): 69 ROS1-Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer patients will be enrolled in Arm A and treated with talerectinib
  Interventions: Drug: Taletrectinib
- Crizotinib (Active Comparator): 69 ROS1-Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer patients will be enrolled in Arm B and treated with Crizotinib
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Taletrectinib — Approximately 138 ROS-1TKI- naïve ROS1+NSCLC patients will be randomized in a 1:1 ration to one of 2 study arms: Arm A: Taletrectinib monotherapy at 600 mg once daily (QD), continuously; Arm B: Crizotinib monotherapy at 250 mg twice daily (BID), continuously.
  Each cycle duration will be 28 days. Participants will be treated until they experience progressive disease (PD) assessed by the blinded Independent Review Committee (BIRC), intolerable toxicity, or another discontinuation criterion is met.
  Arms: Taletrectinib
Drug: Crizotinib — Approximately 138 ROS-1TKI- naïve ROS1+NSCLC patients will be randomized in a 1:1 ration to one of 2 study arms: Arm A: Taletrectinib monotherapy at 600 mg once daily (QD), continuously; Arm B: Crizotinib monotherapy at 250 mg twice daily (BID), continuously.
  Each cycle duration will be 28 days. Participants will be treated until they experience progressive disease (PD) assessed by the blinded Independent Review Committee (BIRC), intolerable toxicity, or another discontinuation criterion is met. Crossover from control group (crizotinib) to taletrectinib is also permitted, at the Investigator's discretion with the Sponsor's approval, for qualifying participants who have experienced objective progression confirmed by the BIRC.
  Arms: Crizotinib

SUMMARY:
This is a Phase 3, randomized, open-label, comparative, multicenter, international study for NSCLC patients whose tumor tissue exhibits ROS1 fusion positivity (i.e., ROS1+) and who have not previously received an ROS1-targeted TKI (i.e., ROS1-TKI-naïve).

Approximately 138 ROS-1 TKI- naïve ROS1+NSCLC patients will be randomized in a 1:1 ration to one of 2 study arms:

* Arm A: Taletrectinib monotherapy at 600 mg once daily (QD), continuously;
* Arm B: Crizotinib monotherapy at 250 mg twice daily (BID), continuously. Each cycle duration will be 28 days.

Participants will be stratified by the presence of intracranial metastases at baseline (Yes versus No) and prior chemotherapy use for locally advanced or metastatic disease (Yes versus No). For the purposes of stratification, prior chemotherapy is defined as completion of ≥1 cycle of chemotherapy in the locally advanced or metastatic setting. Participants will be treated until they experience progressive disease (PD) assessed by the BIRC, intolerable toxicity, or another discontinuation criterion is met. Crossover from control group (crizotinib) to taletrectinib is also permitted, at the Investigator's discretion with the Sponsor's approval, for qualifying participants who have experienced objective progression confirmed by the BIRC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of locally advanced or recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC.
2. Have documentation of ROS1 rearrangement by a positive result
3. Have at least 1 measurable (i.e., target) lesion by Investigator assessment per RECIST v1.1.
4. Prior brain or leptomeningeal metastases allowed if asymptomatic and diagnosed incidentally at study baseline. If participants have neurological symptoms or signs due to CNS metastasis, participants need to complete local therapy (surgery and/or radiation) at least 7 days before enrollment and be clinically stable without requiring for an increasing dose of corticosteroids or use of anticonvulsants to control symptoms.
5. Age ≥18 years (or ≥20 years as required by local regulations).
6. Eastern Cooperative Oncology Group (ECOG) performance status zero (0) to 1.
7. Minimum life expectancy of 3 months or more.
8. Adequate organ function meeting the following criteria:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): ≤3.0 × upper limit of normal (ULN) (or ≤5.0 × ULN, for participants with concurrent liver metastases).
   2. Serum total bilirubin: ≤1.5 × ULN (≤3.0 × ULN for participants with Gilbert syndrome).
   3. Absolute neutrophil count: ≥1500/μL.
   4. Platelet count: ≥75,000/μL.
   5. Hemoglobin: ≥9.0 g/dL.
   6. Estimated creatinine clearance (CLcr) ≥45 mL/min as calculated using the method standard for the institution (e.g., Cockcroft-Gault Equation, i.e., CCr={((140-age)×weight)/(72×SCr)}×0.85 (if female) (Cockcroft and Gault 1976).
9. All toxicities from prior anticancer therapy have resolved to ≤ Grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0), or have resolved to previous baseline, at the time of randomization.
10. The participant is willing and capable of giving written informed consent.

Exclusion Criteria:

1. Previously received an investigational antineoplastic agent for NSCLC.
2. Previously received any prior TKI, including ROS1-targeted TKIs.
3. Received immune checkpoint inhibitors for locally advanced or metastatic disease.
4. Previously received more than 1 regimen of systemic anticancer therapy for locally advanced or metastatic disease.
5. Had major surgery within 28 days prior to randomization. Minor surgical procedures, such as catheter placement or minimally invasive biopsy, are allowed.
6. Have symptomatic CNS metastases (parenchymal or leptomeningeal) at Screening or asymptomatic disease requiring an increasing dose of corticosteroids to control symptoms within 7 days prior to randomization. Participants with no prior history of signs or symptoms of CNS metastases but who receive prophylactic steroids or anticonvulsants are allowed.
7. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging). Participants with leptomeningeal disease and without cord compression are allowed.
8. Uncontrolled pleural, abdominal, or pericardial effusion within 28 days prior to randomization, which is associated with malignant effusion requiring recurrent drainage procedures (once monthly or more frequently).
9. Have been diagnosed with another primary malignancy other than NSCLC except for adequately treated nonmelanoma skin cancer or cervical cancer in situ; definitively treated nonmetastatic prostate cancer; or participants with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
10. Have clinically significant cardiovascular diseases within 6 months prior to randomization: myocardial infarction, severe/unstable angina, coronary/peripheral endovascular treatment, heart failure, cerebrovascular disorder including transient ischemic attack, pulmonary embolism, deep venous thrombosis and or other clinically significant thrombosis.
11. Have a known history of uncontrolled hypertension. Participants with hypertension should be under treatment on study entry to control blood pressure.
12. Have ongoing cardiac dysrhythmias of ≥CTCAE Grade 2, uncontrolled atrial fibrillation of any grade, or QT interval corrected for heart rate by Fredericia's formula (QTcF) >470 milliseconds (female) or >450 milliseconds (male), or symptomatic bradycardia <45 bpm within 6 months before enrollment; participants treated with medications known to be associated with the development of TdP .
13. Have active and clinically significant bacterial, fungal, or viral infection including but not limited to hepatitis B virus (HBV), hepatitis C virus (HCV), known HIV or AIDS-related illness
14. Currently have or have a history of interstitial lung disease (ILD), drug-related pneumonitis, or radiation pneumonitis that required steroid treatment.
15. Be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
PFS (Assessed by BIRC) | About 49 months
  Progression-Free-Survival, The time between the beginning of treatment and the occurrence of disease progression or death. Assessed by the blinded Independent Review Committee (BIRC), per RECIST v1.1

SECONDARY OUTCOMES:
PFS (Assessed by investigator) | About 69months
  Progression-Free-Survival is defined as the time between the beginning of treatment and the occurrence of disease progression or death. Assessed by the investigator, per RECIST v1.1 criteria.
ORR | About 69 months
  Proportion of subjects with the best overall confirmed response of complete response (CR) or partial response (PR) according to RECIST v1.1 criteria.
DOR | About 69 months
  Defined as the time from the first date of objective response (CR or PR) to the first documented date of disease progression. Response assessments are per RECIST v1.1 criteria.
DCR | About 69 months
  Defined as the proportion of subjects with a best overall response of CR, PR or stable disease per RECIST v1.1 criteria) as assessed by the investigator
TTR | About 69 months
  Defined as the overall time from the time of tumor occurrence to the patient's death. Response assessments are per RECIST v1.1 criteria.
OS | About 69 months
  Defined as the time from the first dose to death due to any cause.
IC-TTP | About 69 months
  Defined as the overall time from the time of tumor occurrence with CNS(central nervous system) metastases to the patient's death, Assessed by the BIRC, per RECIST v1.1 criteria.
IC-ORR | About 69 months
  Proportion of CNS metastatic subjects with the best overall confirmed response of complete response (CR) or partial response (PR), Assessed by the BIRC, per RECIST v1.1 criteria.
IC-DOR | About 69 months
  Defined as the time from the first date of objective response (CR or PR) to the first documented date of disease progression on CNS metastatic subjects. Assessed by the BIRC, per RECIST v1.1 criteria.
IC-PFS | About 69 months
  Defined as the time between the beginning of treatment and the occurrence of disease progression or death on CNS metastatic subjects, Assessed by the BIRC, per RECIST v1.1 criteria
IC-PR at 6, 12, 18, 24, and 36 months | About 69 months
  Partial response at 6, 12, 18, 24, and 36 months on CNS metastatic subjects, Assessed by the BIRC, per RECIST v1.1 criteria.
AE | About 69 months
  Adverse event, including the events reported following physical examination, vital signs assessment, clinical laboratory assessment or electrocardiogram(ECG)
Taletrectinib concentration in plasma | About 12 months, at the begining of cycle 1, cycle 2, cycle 7 and cycle 12（each cycle is 28 days）
  Defined as the relationship between taletrectinib concentration and time in the body
patient-reported outcomes(PRO) assessed by EORTC QLQ-C30 | About 69 months
  Patient-reported outcomes of health-related quality of life, assessed by EORTC QLQ-C30, the single-item measures range in score from 0 to 4 or 7, a high score for a symptom scale represents a high level of symptomatology / problems.
PRO assessed by EORTC QLQ-L13 | About 69 months
  Patient-reported outcomes of health-related quality of life, assessed by EORTC QLQ-LC13, the single-item measures range in score from 0 to 4, a high score for a symptom scale represents a high level of symptomatology / problems.
PRO assessed by EQ-5D-5L | About 69 months
  Patient-reported outcomes of health-related quality of life, assessed by EQ-5D-5L, the scale measures range in score from 0 to 100, a high score for the health status represents a high quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai East Hospital
Locations (29):
- China (29):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Linyi Cancer Hospital, Linyi, Shandong
  - Cancer Hospital of Shandong First Medical University, Jinan, Shangdong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang